CLINICAL TRIAL: NCT03029793
Title: Combination of Molecular Biomarkers and Functional Imaging in Predicting Pathologic Response and Clinical Outcomes in Squamous Esophageal Cancer Patients Who Undergo Trimodality Therapy
Brief Title: Biomarkers and Functional Imaging in Predicting Response of Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, Professor, Air Force Military Medical University, China
Other Study IDs: XJFL-2016-ESO
Record Dates: First submitted 2017-01-05; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Prediction; Biomarker; MRI-DWI; PET-CT
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarkers and Imaging analysis: This study will prospectively collect the tissue and blood samples of locally advanced esophageal cancer patients, perform CRT resistance biomarkers testing and functional imaging analysis including SUV value and texture parameters of 18F-FDG PET-CT as well as ADC values DWI-MRI before treatment, 2-3 weeks after the initiation of CRT, and 4 weeks post-nCRT. The investigators will use advanced statistical tools to establish the model and further validate the model in another group of patients. The investigators will also establish a model for survival prediction.
  Interventions: Other: Biomarkers Testing; Other: Functional Imaging analysis

INTERVENTIONS:
Other: Biomarkers Testing — CRT resistance biomarkers will be detected before CRT, 2-3 weeks after the initiation of CRT, and 4 weeks post-CRT.
Other: Functional Imaging analysis — The SUV value and texture parameters of 18F-FDG PET-CT as well as ADC values DWI-MRI will be measures before CRT, 2-3 weeks after the initiation of CRT, and 4 weeks post-CRT.

SUMMARY:
The purpose of this study is to determine whether combination of molecular and biomarkers with functional imaging can predict pathologic response and clinical outcomes in squamous esophageal cancer patients who undergo trimodality therapy which includes neoadjuvant chemoradiotherapy and surgery

DETAILED DESCRIPTION:
The recommended care for the management of locally advanced esophageal cancers is neoadjuvant chemoradiotherapy (nCRT) followed by esophagectomy based on the NCCN guideline. The rate of pathologic complete response (pCR) after nCRT was around 25-30%, reflecting potential cure of unresectable esophageal cancer receiving CRT. Since esophagectomy might have substantial morbidity and mortality rate, establishing the model for predicting nCRT response and survival will guide neoadjuvant treatment decisions and personalized treatment. Thus surgery might be spared in some patients with complete responses after nCRT, and surgery could be selectively reserved for those with only partial or no response to CRT. However, reported models yield unsatisfactory results due to small sample size and low accuracy, and most cases were adenocarcinoma and few models were used to predict survival. This study will prospectively collect the tissue and blood samples of locally advanced esophageal cancer patients, detect CRT resistance biomarkers, assess the SUV value and texture parameters of 18F-FDG PET-CT as well as ADC values DWI-MRI. The investigators will use advanced statistical tools to establish the model and further validate the model in another group of patients.The investigators will also establish a model for survival prediction. This model might possibly guide the personalized treatment for esophageal squamous cell carcinoma patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologic documentation of squamous carcinoma of the esophagus at Xijing Hospital.
2. Newly diagnosed Patients with localized carcinoma of the esophagus who have undergone standard testing and been evaluated by the multidisciplinary team at Xijing Hospital and are considered appropriate candidates for and are willing to undergo chemoradiotherapy followed by surgery at Xijing Hospital.
3. Patient must have undergone a baseline esophageal-gastroduodenoscopy (EGD) with biopsy and endoscopic ultrasonography at Xijing, with tissue available for biomarker analysis.
4. Patient must be willing to undergo this research and must provide written informed consent.

Exclusion Criteria:

1. Patient is unable or unwilling to comply with the requirements of the protocol.
2. History of prior malignancy within the past 3 years.
3. Patients with second primary tumors.
4. Patients who received endoscopical therapy or induction chemotherapy prior to chemoradiation therapy are excluded.
5. Patient is not a candidate for chemoradiation followed by surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with localized carcinoma of the esophagus
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Response | Approximately 12 months
  Mandard tumor regression grade (TRG) was used for pathology analysis. Primary tumor and positive lymph node regression were classified into five histologic tumor regression grades. Grade 1 (complete regression) showed absence of histologically identifiable residual cancer and fibrosis extending through the different layers of the esophageal wall, with or without granuloma. Grade 2 was characterized by the presence of rare residual cancer cells scattered through the fibrosis. Grade 3 involved an increase in the number of residual cancer cells, but fibrosis still predominated. Grade 4 showed residual cancer outgrowing fibrosis. Grade 5 was characterized by the absence of regressive changes.

SECONDARY OUTCOMES:
Overall Survival | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Mei Shi, MD, Study Chair — Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No